CLINICAL TRIAL: NCT07266701
Title: Precision Implant Dentistry - Bite Force Registration as Risk Assessment in Dental Implant Treatment.
Brief Title: The General Aim is to Implement Clinical Assessment of Overload by Voluntary Bite Force Registration to Enable Future Simple But Precise Risk Assessment to Provide Individualized Treatment Plans.
Acronym: Bite force
Status: Enrolling by invitation | Type: Observational
Sponsor: Malmö University (Other)
Collaborators: Smile Tandvård (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-00618-01
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant; Bruxism; Bite Force; Dental Prosthesis Complication; Overload
Keywords: Dental implant; Bite force; dental prosthetic complications; overload
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults 18 - 75 years and above who will undergo a dental implant treatment
  Interventions: Diagnostic Test: Bite force device. Innobyte Kube Innovation TM; Radiation: dental radiology

INTERVENTIONS:
Diagnostic Test: Bite force device. Innobyte Kube Innovation TM — The study is not really an intervention
Radiation: dental radiology — It is a routine modality to take xray to se implant connection and marginal bone level.

SUMMARY:
The general aim of this clinical trial is to implement clinical assessment of overload by bite force registration to enable future simple but precise risk assessment to provide individualized treatment plans.

The main questions it aims to answer are:

* Can we risk-assess patients regarding overload based on bite force measurement before dental implant treatment?
* Can we profile patients based on bite force to tailor precise dental implant treatment for individual patients?
* Will this profiling lead to improved prognosis by reduced number of technical and/or biological complications?

Participants with dental implant prostheses get their bite force measured and followed every year up to 10 years to see complications.

DETAILED DESCRIPTION:
The general aims will be tried to answer with two studies. One prospect and one retrospective.

Specific research questions - Study 2: Prospective clinical trial analyzing bite force and technical complications in patients receiving dental implant treatment.,

* Does bite force differ between patients who do/do not experience complications?
* Does high bite force measurement correlate with the number of technical complications in patients receiving dental implant treatment in a normal population?
* Can we identify at what force risk for fractures becomes significant?
* Does high bite force correlate with peri-implant bone loss?

Patients who accept participation will attend an examination where bilateral bite force will be recorded usin Innobyte, a highly sensitive, calibrated bilateral transducer (InnobyteTM, Kube Innovation) capable of measuring wide ranges of bite forces with good accuracy using digital display not visible to the participant.

Experimental procedure Participants are instructed to abstain from using analgesics or alcohol for 24 hours before the test as well as eating, chewing gum or tobacco products 1 hour before the session.

Participants will be seated upright in a dental chair. Participants will perform one initial maximum bite force registration to familiarize themselves with the equipment. After this, the participants will be asked to bite on the padded force transducer as hard as possible (the time needed to achieve maximum bite force is determined by the subject but typically 2 to 5 seconds). Three such measurements will be recorded with a 30-second rest in between, and the average will be calculated and registered.

All tests are carried out in one experimental session that will take approximately 10 minutes.

Baseline radiographs as well as radiographs taken at follow-up visits will be reviewed for signs of bone loss. Registrations of bleeding on probing and pocket depth will be done to determine presence of peri-implant mucositis or peri-implantitis.

Any identified technical or biological complications and/or signs of wear (measured according to TWES 3.0) will be registered together with data regarding patient age and gender, type of implant restoration, restorative material, opposing dentition and time after delivery of the prosthetic construction.

Participants will be asked to answer a questionnaire evaluating orofacial pain and jaw function and factors that may affect this. The questionnaire includes initial screening questions as well as validated instruments:

* Screening - 3Q/TMD
* Stress - PSS-10
* Jaw function - JFLS-8
* Use of splint
* Brux-Screen

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above that understand written and spoken Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients who are planned to undergo, or who have undergone, dental implant treatment at any of the general dentist clinics within the Smile Tandvård AB group and other private practices and university setting at Malmö University, Universitetstandvården.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2035-05-15 (Estimated)

PRIMARY OUTCOMES:
Bite force in correlation to technical and biological complications in patients with dental implant treatment | 2025-2028

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bergengren, Study Chair — Malmö University Dental school
Locations (1):
- Malmö University, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No